CLINICAL TRIAL: NCT00293527
Title: A Phase II Dose Escalation Study of Continuous Daily Subcutaneous Administration of Interferon Alpha-2b in Patients With Metastatic or Unresectable Clear Cell Renal Cell Carcinoma
Brief Title: Interferon Alpha-2b (Intron A) for Metastatic or Unresectable Clear Cell Renal Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn in October 2006, no longer of interest
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Thomas Olencki, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-05030
Record Dates: First submitted 2006-02-15; First posted 2006-02-17 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Renal Cancer
Keywords: Metastatic
MeSH Terms: conditions — Kidney Neoplasms; Neoplasm Metastasis | interventions — Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Interferon Alpha-2b

SUMMARY:
This study will determine the response rate of daily low dose interferon-alpha-2b in patients with metastatic or unresectable clear cell renal cell carcinoma.

DETAILED DESCRIPTION:
Rationale: Interferon has long been used as a therapy for renal cell carcinoma. However, optimal dosing schedules have not been identified and patients have been relegated to receiving the highest possible doses for prolonged periods of time. This high-dose approach often leads to serious adverse effects from toxicity that limits the usefulness and patient tolerance of this treatment. No formal study has determined the relationship if any between the maximal tolerated dose (MTD) and the biological effective dose of interferon alpha-2b. The current study seeks to fill that gap by gathering research information about different doses of interferon alpha-2b and correlating with measurements of JAK/STAT in the blood. Validation of correlative studies to determine optimum biologic dosing are needed so that therapy may be adjusted appropriately rather then the current approach of maximizing dose. In addition, a trial of low dose daily administered interferon-2b has not been carried out in the current era with refined histologic classification and modern CT imaging scanning. As this therapy potentially has wide applicability, definite response rates need to be documented.

Purpose: The purpose of this study is to assess the response rate of daily low dose interferon-2b in patients with metastatic or unresectable clear cell renal carcinoma. The duration of the response and overall survival will be determined in study participants. This study will also evaluate JAK/STAT, two types of kinases or enzymes involved in an intracellular signaling process associated with cancer growth, in peripheral blood mononuclear cells over the course of interferon alpha-2b dose escalation. Researchers will examine in a preliminary manner the correlation between clinical response, toxicity, and JAK/STAT signal transduction. Progression free survival and rate of stable disease will also be determined in a preliminary manner.

Treatment: Study participants will receive interferon alpha-2b. This drug will be self-administered daily through injections into the skin. The dose level of interferon alpha-2b will be increased each week into study treatments. For the first three weeks and approximately monthly thereafter, patients will have blood drawn three hours following interferon alpha-2b administration to measure JAK/STAT. Toxicity from study treatments will be closely monitored in patients during clinics visits. Supportive care therapies will be given throughout the study. Treatments will be discontinued due to disease growth or unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or unresectable clear cell renal cell carcinoma
* Measurable disease

Exclusion Criteria:

* Prior interferon therapy
* More than 3 prior therapy regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Olencki, Principal Investigator — Ohio State University